CLINICAL TRIAL: NCT06559553
Title: A Prospective Clinical Study of "Selinexor+Pegaspargase+Dexamethasone" in the Treatment of Stage Ⅰ/Ⅱ NK/ T-Cell Lymphoma
Brief Title: "Selinexor+Pegaspargase+Dexamethasone"in Ⅰ/Ⅱ NKTCL
Acronym: Selinexor
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mingzhi Zhang (Other)
Responsible Party: Sponsor-Investigator, Mingzhi Zhang, the director of oncology department of the first affiliated hospital, Zhengzhou University
Organization: Zhengzhou University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: hnslblzlzx202207
Record Dates: First submitted 2024-08-15; First posted 2024-08-19 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: NKTCL; Selinexor
Keywords: NKTCL; Selinexor

STUDY DESIGN:
Intervention Model Description: Climbing stage, and the following two stages of research
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Selinexor+pegaspargase+dexamethasone (Experimental): Nuclear export protein-1 is the main transporter protein for leucine-rich proteins to enter the cytoplasm from the nucleus through the nuclear pore complex, which is overexpressed in malignant tumor cells. Studies have shown that Selinexor inhibits the nuclear export of viral mRNA such as EBV, and has good therapeutic potential for NKTCL. Selinexor combined with pemaspartase, dexamethasone and sequential radiotherapy may be the golden choice for early NK/T cell lymphoma, improving the local control rate of the disease and improving the overall prognosis of NK/T cell lymphoma.
  Interventions: Drug: Selinexor+pegaspargase+dexamethasone

INTERVENTIONS:
Drug: Selinexor+pegaspargase+dexamethasone — Nuclear export protein-1 is the main transporter protein for leucine-rich proteins to enter the cytoplasm from the nucleus through the nuclear pore complex, which is overexpressed in malignant tumor cells. Studies have shown that Selinexor inhibits the nuclear export of viral mRNA such as EBV, and has good therapeutic potential for NKTCL. Selinexor combined with pemaspartase, dexamethasone and sequential radiotherapy may be the golden choice for early NK/T cell lymphoma, improving the local control rate of the disease and improving the overall prognosis of NK/T cell lymphoma.

SUMMARY:
evaluate the efficacy and safety of "Selinexor+pegaspargase+dexamethasone" in early stage NK/ T-cell lymphoma

DETAILED DESCRIPTION:
Patients with early NK/T cell lymphoma were treated with an oral regimen of "Selinisol + pemaspartase + dexamethasone"

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years old, ECOG score 0-2; (including those aged 18 and 70);
2. Pre-survival time > 6 months;
3. The pathological tissue was confirmed as NK/T cell lymphoma (the pathological report of the first three months of enrollment could be accepted) (Note: If there is any doubt about the pathological diagnosis, domestic third-party consultation could be organized);
4. Clinical stage Ⅰ to Ⅱ (CA stage) with at least one measurable lesion;
5. Acceptable hematological indicators, no contraindications to chemotherapy; Neutrophil absolute value ≥1.0×10^9 /L, platelet ≥75×10^9 /L, hemoglobin ≥80g/L (except patients with lymphoma bone marrow infiltration);
6. Liver function: direct bilirubin ≤1.5× upper limit reference value; Glutamic pyruvic transaminase or glutamic oxalacetic transaminase ≤2.5× upper limit reference value; Alkaline phosphatase ≤3×ULN in non-bone invaded patients;
7. Renal function: serum creatinine ≤1.5×ULN;
8. Female and male patients of reproductive age and their spouses are willing to use adequate contraception throughout the study period, and female patients of reproductive age must have a negative serum pregnancy test within 7 days before the first dose;
9. The newly treated patient had not received other tumor-related treatment in the past;
10. Subjects voluntarily participate in the clinical trial, sign informed consent, and cooperate with follow-up;

Exclusion Criteria:

1. Refuse to collect blood samples;
2. Previous allergy to any of the drugs in the program;
3. Pregnant and lactating women;
4. Major diseases that the investigator believes can cause interference with the test;
5. Combined with other tumors;
6. There are contraindications related to therapeutic drugs in the program;
7. Persons with serious mental illness;
8. Participating in other clinical trials;
9. Previous anti-tumor therapy (such as radiotherapy, chemotherapy, hormone therapy, biotherapy, immunotherapy);
10. Other serious medical conditions that may limit participants' participation in the trial, such as uncontrolled diabetes; Severe cardiac insufficiency (NYHA grade II or above); Acute coronary syndrome within the last 6 months; Coronary revascularization such as stenting, coronary artery bypass surgery, and other heart and large vessel related procedures within the last 6 months; Severe arrhythmias include frequent ventricular early, ventricular tachycardia, rapid atrial fibrillation/flutter, and severe bradycardia. Uncontrolled hypertension: systolic blood pressure >150mmHg, diastolic blood pressure >100mmHg. Gastric ulcers (stomach ulcers that researchers have determined are at risk of perforation); Active autoimmune diseases (e.g. systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, Sjogren's syndrome, autoimmune thrombocytopenia, etc.); Severe respiratory disease (such as obstructive pulmonary disease and a history of bronchospasm);
11. Hemophagic cell syndrome;
12. Researchers do not consider it suitable for inclusion;
13. Hepatitis B core antibody (HBcAb) positive and peripheral blood hepatitis B virus (HBV) DNA titer detection is not within the normal reference value range; Hepatitis C virus (HCV) antibody positive and peripheral blood hepatitis C virus (HCV) RNA positive; Human immunodeficiency virus (HIV) antibody positive; Syphilis test positive.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
CRR | From date of randomization until the date tumor volume has reduced, assessed up to 36 months
  The proportion of patients whose tumor volume has reduced to a predetermined value and can maintain the minimum time limit is the sum of complete mitigation.

CONTACTS AND LOCATIONS:
Locations (1):
- Oncology Department of The First Affilliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No